CLINICAL TRIAL: NCT07190690
Title: Comparison of a Contemporary Sirolimus-eluting Stent (ihtDEStiny®) With Another Everolimus-eluting Stent (Xience™), Both With Permanent Polymers, in Patients With Acute Coronary Syndrome and de Novo Coronary Artery Lesions (DestinACSion Study)
Brief Title: Comparison of a Contemporary Sirolimus-eluting Stent (ihtDEStiny®) With Another Everolimus-eluting Stent (Xience™), Both With Permanent Polymers, in Patients With Acute Coronary Syndrome and de Novo Coronary Artery Lesions
Acronym: DestinACSion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC45-DestinACSion
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: Drug Eluting Stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator: ihtDEStiny® DES (Other)
  Interventions: Device: ihtDEStiny® DES implanted
- Experimental: Xience™ DES (Other)
  Interventions: Device: Xience™ DES implanted

INTERVENTIONS:
Device: ihtDEStiny® DES implanted — ihtDEStiny® DES implanted
  Arms: Active Comparator: ihtDEStiny® DES
Device: Xience™ DES implanted — Xience™ DES implanted
  Arms: Experimental: Xience™ DES

SUMMARY:
To evaluate the efficacy of the two DES (Drug Eluting Stent) used in terms of device-related adverse events at 12 months after PCI (Percutaneous Coronary Intervention).

To compare the clinical safety and efficacy by comparing net clinical events (defined as the combination of ischemic and hemorrhagic events) of the two DES used at 12 months after PCI.

DETAILED DESCRIPTION:
To evaluate the efficacy of the two DES (Drug Eluting Stent) used in terms of device-related adverse events at 12 months after PCI (Percutaneous Coronary Intervention).

To compare the clinical safety and efficacy by comparing net clinical events (defined as the combination of ischemic and hemorrhagic events) of the two DES used at 12 months after PCI.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet ALL inclusion criteria will be included:

* Patients aged ≥18 years, and
* Patients diagnosed with an acute coronary syndrome (ACS), either SCASEST (Acute Coronary Syndrome without Persistent ST-Segment Elevation) or IAMCEST (Acute Myocardial Infarction with Persistent ST-Segment Elevation), for which they will undergo PCI, and
* Patients with de novo lesions in vessels with a reference diameter of ≥2.25 mm and ≤4.5 mm in whom implantation of one or more DES is clinically indicated, and
* Patients who have been informed of the characteristics of the study and have provided written informed consent.

Exclusion Criteria:

Patients must not meet any of the following exclusion criteria:

* Patients in cardiogenic shock according to the severity criteria defined by the Society of Cardiovascular Angiography and Interventions (SCAI): "C" (Classic Shock), "D" (Deteriorating) and "E" (Extremis).
* Patients unable to provide informed consent.
* Patients with a known hypersensitivity or allergy to aspirin or any P2Y12 receptor inhibitor (clopidogrel, prasugrel, ticagrelor), heparin, contrast agents, or any of the components of DES.
* Patients with active bleeding at the time of PCI requiring medical attention.
* Patients with planned surgery within the next 3 months.
* Patients with any medical condition that limits a life expectancy of less than 12 months.
* Patients participating in another clinical trial in which the primary endpoint was not met.
* Pregnant or breastfeeding women of childbearing potential with a positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2029-10-15 (Estimated); Study Completion 2030-10-15 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: Device-oriented Composite Endpoint (DoCE) | 12 months
  Composite clinical endpoint cardiac Rate at 12 months cause death, target vessel myocardial infraction (TV-MI), and Clinically individual target lesion revascularization (CI-TLR)
NACE | 12 months
  Composite clinical endpoint Rate of all-cause death, any stroke, any MI, any revascularization and BARC type 3 or 5 bleeding events

SECONDARY OUTCOMES:
All-Cause Death Rate at 12 months | 12 months
  All-Cause Death Rate at 12 months
All-Cause Death Rate at 24 months | 12 months
  All-Cause Death Rate at 24 months
Cardiac Death Rate at 12 months | 12 months
  Cardiac Death Rate at 12 months
Cardiac Death Rate at 24 months | 12 months
  Cardiac Death Rate at 24 months
Myocardial Infarction Rate at 12 months | 12 months
  Myocardial Infarction Rate at 12 months
Myocardial Infarction Rate at 24 months | 12 months
  Myocardial Infarction Rate at 24 months
Periprocedural myocardial infarction Rate | PCI procedure
  Periprocedural myocardial infarction Rate
Definite/Probable stent thrombosis rate at 12 months | 12 months
  Definite/Probable stent thrombosis rate at 12 months
Definite/Probable stent thrombosis rate at 24 months | 24 months
  Definite/Probable stent thrombosis rate at 24 months
Any stroke at 12 months | 12 months
  Stroke Rate at 12 months
Any stroke at 24 months | 12 months
  Stroke Rate at 24 months
BARC type 2 ,3 or 5 bleeding events at 12 months | 12 months
  Bleeding events type 2, 3 or 5 defined by BARC (Bleeding Academic Research Consortium) criteria at 12 months
BARC type 2 ,3 or 5 bleeding events at 24 months | 24 months
  Bleeding events type 2, 3 or 5 defined by BARC (Bleeding Academic Research Consortium) criteria at 24 months
Target vessel revascularization Rate at 12 months | 12 months
  Target vessel revascularization Rate at 12 months
Target vessel revascularization Rate at 24 months | 24 months
  Target vessel revascularization Rate at 24 months
Target vessel Failure (TVF) Rate at 12 months | 12 months
  Target vessel Failure (TVF) Rate at 12 months
Target vessel Failure (TVF) Rate at 24 months | 24 months
  Target vessel Failure (TVF) Rate at 24 months
Target Lesion Failure (TLF) Rate at 12 months | 12 months
  Target Lesion Failure (TLF) Rate at 12 months
Target Lesion Failure (TLF) Rate at 24 months | 24 months
  Target Lesion Failure (TLF) Rate at 24 months
Target Vessel Revascularization Rate (TVR) at 12 months | 12 months
  Target Vessel Revascularization Rate (TVR) at 12 months
Target Vessel Revascularization Rate (TVR) at 24 months | 24 months
  Target Vessel Revascularization Rate (TVR) at 24 months
Target lesion ischemia-guided revascularization Rate at 12 months | 12 months
  Target lesion ischemia-guided revascularization Rate at 12 months
Target lesion ischemia-guided revascularization Rate at 24 months | 24 months
  Target lesion ischemia-guided revascularization Rate at 24 months
Repeated revascularization Rate at 12 months | 12 months
  Repeated revascularization Rate at 12 months
Repeated revascularization Rate at 24 months | 24 months
  Repeated revascularization Rate at 24 months
Major Adverse Cardiac Events (MACE) Rate at 12 months | 12 months
  Major Adverse Cardiac Events (MACE) Rate is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization at 12 months
Major Adverse Cardiac Events (MACE) Rate at 24 months | 24 months
  Major Adverse Cardiac Events (MACE) Rate is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization at 24 months

CONTACTS AND LOCATIONS:
Locations (7):
- Spain (7):
  - Hospital Universitario San Juan Alicante, Alicante
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Universitario de Leon, León
  - Hospital Universitario Lucus Agustí, Lugo
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Background] de la Torre Hernandez JM, Otaegui I, Subinas A, Gomez-Menchero A, Moreno R, Rondan J, Munoz-Garcia E, Sainz-Laso F, Garcia Del Blanco B, Rumoroso JR, Diaz JF, Berenguer A, Gomez-Lara J, Zueco J. First-in-Man Evaluation of a Sirolimus-Eluting Stent With Abluminal Fluoropolymeric/Triflusal Coating With Ultrathin Struts by OCT at 9 Months' Follow-Up: The PROMETHEUS Study. Cardiovasc Revasc Med. 2021 Nov;32:18-24. doi: 10.1016/j.carrev.2020.12.025. Epub 2020 Dec 29. PMID 33386256
- [Background] Ploumen EH, von Birgelen C. Novel DES Aims at Full Thromboresistance: Another Promising Player on the Field? Cardiovasc Revasc Med. 2021 Nov;32:25-26. doi: 10.1016/j.carrev.2021.07.029. Epub 2021 Aug 11. No abstract available. PMID 34391680
- [Background] Linares Vicente JA, Sainz Laso F, Casanova Sandoval JM, Rumoroso Cueva JR, Gomez Menchero A, Gomez Hospital JA, Perez Guerrero A, Santos Martinez S, Fernandez Portales J, Romani S, Garcia Del Blanco B, Ocaranza Sanchez R, Urbano Carrillo C, Garcia San Roman K, Vinhas H, Cid Alvarez B, Sanchis Fores J, Telleria Arrieta M, Torres Bosco A, Pinar Bermudez E, Mendez Castro JJ, Lozano Ruiz de Poveda F, Perez de Prado A, De la Torre Hernandez JM. Long-term outcomes of hydrodynamic ultra-thin strut sirolimus-eluting stent with fluoropolymer containing triflusal: VELAZQUEZ-EPIC26 study. Cardiovasc Revasc Med. 2025 Jul 17:S1553-8389(25)00392-6. doi: 10.1016/j.carrev.2025.07.009. Online ahead of print. PMID 40713212
- [Background] Zaman A, de Winter RJ, Kogame N, Chang CC, Modolo R, Spitzer E, Tonino P, Hofma S, Zurakowski A, Smits PC, Prokopczuk J, Moreno R, Choudhury A, Petrov I, Cequier A, Kukreja N, Hoye A, Iniguez A, Ungi I, Serra A, Gil RJ, Walsh S, Tonev G, Mathur A, Merkely B, Colombo A, Ijsselmuiden S, Soliman O, Kaul U, Onuma Y, Serruys PW; TALENT trial investigators. Safety and efficacy of a sirolimus-eluting coronary stent with ultra-thin strut for treatment of atherosclerotic lesions (TALENT): a prospective multicentre randomised controlled trial. Lancet. 2019 Mar 9;393(10175):987-997. doi: 10.1016/S0140-6736(18)32467-X. Epub 2019 Feb 28. PMID 30827782
- [Background] Garcia-Garcia HM, McFadden EP, Farb A, Mehran R, Stone GW, Spertus J, Onuma Y, Morel MA, van Es GA, Zuckerman B, Fearon WF, Taggart D, Kappetein AP, Krucoff MW, Vranckx P, Windecker S, Cutlip D, Serruys PW; Academic Research Consortium. Standardized End Point Definitions for Coronary Intervention Trials: The Academic Research Consortium-2 Consensus Document. Circulation. 2018 Jun 12;137(24):2635-2650. doi: 10.1161/CIRCULATIONAHA.117.029289. PMID 29891620